CLINICAL TRIAL: NCT05302505
Title: Impact of Simulation-based Training in Addition to Theoretical Training Versus Theoretical Training Alone for Nurses on the Occurring of Adverse Events Related to Arteriovenous Fistula Puncture in Chronic Hemodialysis Patients.
Brief Title: Simulation-based Training for Nurses and Arteriovenous Fistula Puncture in Chronic Hemodialysis Patients
Acronym: SIMFAV2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2021-A01813-38
Record Dates: First submitted 2022-03-02; First posted 2022-03-31 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Nursing Caries; Arteriovenous Fistula; Simulation-based Training
MeSH Terms: conditions — Arteriovenous Fistula

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Simulation (Experimental): Theoretical training in e-learning for nurses on :
  * arteriovenous fistula puncture
  * use of ultrasound with echoreferencing and ultrasound guidance
  * therapeutic communication
  And simulation-based training (procedural) on :
  * arteriovenous fistula puncture
  * use of ultrasound with echoreferencing and ultrasound guidance
  * therapeutic communication
  Interventions: Other: simulation-based training
- Control (No Intervention): Theoretical training for nurses in e-learning on :
  * arteriovenous fistula puncture
  * use of ultrasound with echoreferencing and ultrasound guidance
  * therapeutic communication

INTERVENTIONS:
Other: simulation-based training — Based-simulation training for nurses in a simulation center : puncture of arteriovenous fistula and utilization of echograph and conversational hypnosis
  Arms: Simulation

SUMMARY:
Currently, the technique of arteriovenous fistula puncture is transmitted by companionship within hemodialysis units. Although the main principles of the technique are well known and common to all hemodialysis units, strong rationales are still lacking to standardize fine practices such as the relative position of the needles, the angle of attack of the needle at puncture, the position of the bevel at the time of puncture and once the needle is in the vascular lumen.

The training of professionals using a simulation-based training program on the approach to arteriovenous fistula puncture, in a process of optimizing practices and continuous improvement of care, while respecting the principles of andragogy, seems to be a suitable tool. This program is built in a multi-professional team from nephrology, nursing and health simulation.

DETAILED DESCRIPTION:
Currently, the technique of arteriovenous fistula puncture is transmitted by companionship within hemodialysis units. Although the main principles of the technique are well known and common to all hemodialysis units, strong rationales are still lacking to standardize fine practices such as the relative position of the needles, the angle of attack of the needle at puncture, the position of the bevel at the time of puncture and once the needle is in the vascular lumen.

The training of professionals using a simulation-based training program on the approach to arteriovenous fistula puncture, in a process of optimizing practices and continuous improvement of care, while respecting the principles of andragogy, seems to be a suitable tool. This program is built in a multi-professional team from nephrology, nursing and health simulation.

The aim of this study is to evaluate whether a simulation-based training program for nurses, concerning arteriovenous fistula puncture puncture, would allow to decrease the adverse events related to punctures.

The investigators propose a prospective, comparative, randomized, multicenter study involving 8 hemodialysis centers. The primary objective is to compare the number of arteriovenous fistula puncture-related adverse events between:

* A group receiving theoretical training + simulation-based training (4 centers)
* A group receiving theoretical training only (4 centers)

Will be included all adult patients who are to receive an arteriovenous fistula puncture puncture by a hemodialysis-trained IDE, during a scheduled chronic dialysis session.

This study is innovative for several reasons:

* simulation-based training in continuing education, among professionals is not widely used
* simulation-based training in continuing education allows the conceptualization of the team approach to VF by its modeling in simulation
* the evaluation of the direct benefit of the training on the patient, a Kirkpatrick level 4, is very little described in the literature.

Thus, this study is of major interest to patients managed in nephrology with the simulation-based training tool.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients
* Arteriovenous fistula puncture in the hemodialysis unit of the nephrology, dialysis, transplantation department
* Nurses trained in hemodialysis

Exclusion Criteria:

* arteriovenous fistula puncture in the emergency area/foldout of the unit
* Refuse of data collection
* Not speak French
* Minor
* Under guardianship or unable to give informed consent
* Not enrolled in a social security plan
* Pregnant or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9600 (Estimated)
Dates: Start 2022-09-05 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Number of adverse events occurring during arteriovenous fistula puncture (comparison of the percentages of event occurrence) | 45 days
  defined by one of the following events:
  * Unipuncture failure
  * Bipuncture failure
  * Simple hematoma
  * Hematoma not allowing continued dialysis

CONTACTS AND LOCATIONS:
Overall Officials: Erwan Guillouët, Principal Investigator — University Hospital, Caen
Locations (9):
- France (9):
  - Center hospital of Alençon, Alençon
  - University hospital center of Caen, Caen
  - Private Hospital St Martin, Caen
  - Center Hospital of Dieppe, Dieppe
  - Center Hospital of Flers, Flers
  - ANIDER, Hérouville-Saint-Clair
  - Center Hospital of Lisieux, Lisieux
  - Anider Alencon, Saint-Germain-du-Corbéis
  - Center Hospital of Memorial United States of St Lo, Saint-Lô

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Guillouet E, Tomadesso C, Flores BA, Henri P, Lanot A, Morello R, Guillouet S. Impact of simulation-based training in addition to theoretical training versus theoretical training of nurses alone in the occurrence of adverse events related to arteriovenous fistula puncture in chronic hemodialysis patients: study for a cluster randomized controlled trial (SIMFAV2). Trials. 2023 Aug 7;24(1):500. doi: 10.1186/s13063-023-07513-8. PMID 37550740